CLINICAL TRIAL: NCT04713722
Title: Early Life Stress and Depression: Molecular and Functional Imaging
Acronym: ELS
Status: Recruiting | Type: Observational
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Diego Pizzagalli, Professor, Harvard Medical School; Director, Mclean Hospital
Other Study IDs: 2020P001470
Record Dates: First submitted 2021-01-14; First posted 2021-01-19 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Depression; Trauma, Psychological
MeSH Terms: conditions — Depression; Psychological Trauma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Inflammation panel with RNA DNA samples for Peripheral blood mononuclear cells (PBMC) purification
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- MDD/childhood adversity group: subjects with current MDD who experienced childhood adversity
- rMDD/ childhood adversity: subjects with a history of MDD who experienced childhood adversity
- MDD: subjects in a current episode of MDD, with no history of childhood adversity
- Healthy Control: healthy control subjects, with no history of childhood adversity

SUMMARY:
Severe childhood adversity accounts for a large portion of psychiatric illness, and an increased risk for major depressive disorder (MDD). For some individuals, childhood adversity has negative psychological and medical consequences; others preserve mental and physical health despite such experiences (they are resilient). In spite of this, little is known about the neurobiological mechanisms related to childhood adversity, especially oxidative stress abnormalities in the brain. To fill this gap, this study combines functional, structural, and molecular imaging approaches to examine the role of oxidative stress abnormalities related to childhood adversity.

DETAILED DESCRIPTION:
Epidemiological studies have shown that severe childhood adversity explains 32-44% of psychiatric disorders, and is associated with 4.6-fold risk for MDD later in life. In spite of these epidemiological data, the neurobiological underpinnings associated with maladaptive sequelae of severe childhood adversity as well as resilience remain largely unknown.

Preclinical research suggests that early adversity leads to (1) structural abnormalities in brain regions critically implicated in stress regulation; (2) increased oxidative stress; and (3) glutamatergic abnormalities. The current research protocol is designed to prospectively test the contributions of these abnormalities in individuals exposed to severe childhood adversity.

Improving our understanding of neurobiological mechanisms associated with different childhood adversity outcomes is of paramount importance in order to (1) identify individuals at risk for psychopathology and maladaptive behavior, (2) prevent re-victimization, and (3) develop more targeted therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

* Females of all races and ethnic origins
* Ages from 20 to 32
* Right-handed
* Capable of providing written informed consent
* Currently unmedicated. Note that this criterion applies at enrollment only, and subjects will be informed that they can continue to be in the study if they begin a new medication after enrollment.
* Normal or corrected-to-normal vision and hearing
* Fluency in written and spoken English
* Absence of first-degree relatives with a history of a psychotic disorder or psychotic symptoms; (adopted individuals are eligible to participate but we will probe about family history in case such information is available to the adopted subject)

Exclusion Criteria:

* Participants with suicidal ideation where continued study participation is deemed unsafe by the study clinician (these participants will be immediately referred to appropriate clinical treatment)
* Pregnant women, or women of childbearing potential who have a positive result on a urine pregnancy test
* Failure to meet MRI safety requirements including but not limited to any metal implants or prostheses that cannot be removed, or exposure to shrapnel
* Claustrophobia or severe anxiety that might impact participation in neuroimaging
* Injury or movement disorder that may make it difficult to lie still in the scanner
* Any current recreational/illicit drug use as assessed by a urine drug test (covering cocaine, cannabinoids, opiates, amphetamines, methamphetamines, phencyclidine, MDMA, benzodiazepines, methadone, oxycodone, tricyclic antidepressants, and barbiturates)
* Use of drug or herbal supplement for depression (e.g., St. John's Wort or SAMe) of those that could affect stress response
* Use of any medication in the 24 hours prior to the Scanning procedure (including antibiotics, asthma inhalants, pain relievers, antihistamines, or over-the-counter medications).
* Recent use (within 3 weeks) or any medication that affects blood flow or blood pressure, or which is vasodilating/vasoconstricting
* Use of Melatonin within 5 days of the Scanning procedure
* Metformin use in the past 6 months (for either clinical care or as part of research)
* Serious or unstable medical illness, including cardiovascular, hepatic, renal, respiratory, endocrine (hypothyroidism), neurologic, autoimmune disease (such as Lyme, Crohn's), or hematologic disease
* Current infectious illness (either transient or chronic); Current episode of allergic reaction or asthma
* Hemophilia; Diabetes with poor glucose control; History of chronic migraine (> 15 days/mo.); History or current diagnosis of dementia
* History of seizure disorder
* Any history of significant head injury or concussion
* Past/current DSM-5 diagnosis of: OCD, ADHD, schizophrenia, schizoaffective disorder, delusional disorder, psychotic disorders NOS, bipolar disorder, patients with mood congruent or mood incongruent psychotic features, autism or any other pervasive developmental disorder, organic mental disorder, anorexia, binge eating disorder or bulimia (however a history of bulimia or binge eating disorder is allowable if it has been in remission for at least two years)
* History of moderate or severe substance or alcohol use disorder; or, mild substance or alcohol use disorder within the last 12 months (with the exception of cocaine or stimulant abuse, which will lead to automatic exclusion).
* History of ECT
* Patient is clinically unstable, in the judgment of the clinician

Ages: 20 Years to 32 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only female
Study Population: Healthy controls, those with depression (current or remitted), and those with depression and history of childhood adversity
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Immuno-oxidative abnormalities | Baseline
  Redox ratio and glutamate metabolites in the prefrontal cortex

SECONDARY OUTCOMES:
Blood oxygen level dependent (BOLD) activation | Baseline
  Prefrontal cortex activation during a reward task
Blood oxygen level dependent (BOLD) activation in emotional processing | Baseline
  Prefrontal cortex activation during an emotional processing task
Peripheral inflammation | Baseline
  Stress-related pro-inflammatory transcription control pathways

CONTACTS AND LOCATIONS:
Overall Officials: Diego Pizzagalli, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States